CLINICAL TRIAL: NCT02209012
Title: Twelve Month Follow-Up Evaluation of Subjects Participating in DUSA-CP0108 (A Phase 3 Study of Photodynamic Therapy With Levulan Kerastick Topical Solution + Blue Light Versus Topical Solution Vehicle + Blue Light for the Treatment of Actinic Keratoses on the Upper Extremities)
Brief Title: Twelve Month Follow-Up of CP0108
Status: Completed | Type: Observational
Sponsor: DUSA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP0108A
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Solutions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ALA: Subjects who received ALA in CP0108
  Interventions: Drug: Aminolevulinic Acid (ALA); Device: BLU-U Blue Light Photodynamic Therapy Illuminator
- Vehicle: Subjects who received Vehicle in CP0108
  Interventions: Drug: Topical Solution Vehicle; Device: BLU-U Blue Light Photodynamic Therapy Illuminator

INTERVENTIONS:
Drug: Aminolevulinic Acid (ALA) — Levulan PDT given in CP0108
  Other Names: Levulan Kerastick
  Groups: ALA
Drug: Topical Solution Vehicle — Vehicle PDT given in CP0108
  Groups: Vehicle
Device: BLU-U Blue Light Photodynamic Therapy Illuminator — PDT given in CP0108

SUMMARY:
The purpose of this study is to determine the long-term safety and efficacy of Levulan PDT in subjects with multiple actinic keratosis of the upper extremities who received treatment as part of the DUSA CP0108 study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have been enrolled in the DUSA-CP0108 study, completed their assigned treatment and Visit 6 (Week 12).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who were enrolled in the DUSA-CP0108 study, completed their assigned treatment (ALA-PDT or vehicle + blue-light) and Visit 6.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Subject Recurrence Rate | Month 12
  percentage of subjects who had achieved 100% clearance at Visit 6 (Week 12) in CP0108, that have one or more previously treated (as part of CP0108) AK lesion(s) present in the Treatment Area at any visit during CP0108A follow-up
Duration of Response | one year
  the time from Week 12 (in the DUSA-CP0108 study) to the visit at which a previously treated and cleared lesion recurs. If a subject begins or receives treatment for previously cleared AK lesions in the Treatment Area between scheduled visits, the date the treatment started will be the end of treatment response, or, if the start date is unknown, the visit prior to starting the new treatment will be the end of treatment response.
Lesion Recurrence Rate | Month 12
  the proportion of lesions that were CR at Week 12 in CP0108 that are visible or palpable at Visit 10, will be determined for all ALA-PDT treated subjects who have at least one AK designated as "clear" at Week 12 in the DUSA-CP0108 study.
Duration of Lesion Response | one year
  the time from Week 12 (in the DUSA-CP0108 study) to the visit at which the AK lesion recurs for all ALA-PDT treated subjects who have at least one AK designated as "clear" at Week 12 in the DUSA-CP0108 study. If a previously cleared lesion receives treatment between scheduled visits, the date the treatment started will be the end of treatment response for that lesion, or, if the start date is unknown, the visit prior to starting the new treatment will be the end of treatment response.

OTHER OUTCOMES:
Hyperpigmentation | Baseline
  HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Hyperpigmentation | Month 3
  HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Hyperpigmentation | Month 6
  HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Hyperpigmentation | Month 9
  HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Hyperpigmentation | Month 12
  HYPERPIGMENTATION SCALE Grade 0 = No hyperpigmentation Grade 1 = Light hyperpigmentation involving small areas Grade 2 = Moderate hyperpigmentation involving small areas; light hyperpigmentation involving moderate areas Grade 3 = Moderate hyperpigmentation involving moderate sized areas; light hyperpigmentation involving large areas; small areas of marked hyperpigmentation Grade 4 = Marked hyperpigmentation involving moderate or large sized areas
Hypopigmentation | Baseline
  HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation
Hypopigmentation | Month 3
  HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation
Hypopigmentation | Month 6
  HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation
Hypopigmentation | Month 9
  HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation
Hypopigmentation | Month 12
  HYPOPIGMENTATION SCALE Grade 0 = No hypopigmentation Grade 1 = Light hypopigmentation involving small areas Grade 2 = Moderate hypopigmentation involving small areas; light hypopigmentation involving moderate areas Grade 3 = Moderate hypopigmentation involving moderate sized areas; light hypopigmentation involving large areas; small areas of marked hypopigmentation
Erythema | Baseline
  Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Erythema | Month 3
  Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Erythema | Month 6
  Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Erythema | Month 9
  Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Erythema | Month 12
  Erythema Scale - Grade 0 = None Grade 1 = Minimal - barely perceptible erythema Grade 2 = Mild - predominantly minimal erythema (pink) in the treated area with or without a few isolated areas of more intense erythema Grade 3 = Moderate - predominantly moderate erythema (red) in the treated area with or without a few isolated areas of intense erythema (bright red) Grade 4 = Severe - predominantly intense erythema (bright red) in the treated area with or without a few isolated areas of very intense (fiery red) erythema
Edema | Baseline
  EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Edema | Month 3
  EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Edema | Month 6
  EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Edema | Month 9
  EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Edema | Month 12
  EDEMA SCALE Grade 0 = None Grade 1 = Minimal - scant, rare edema Grade 2 = Mild - easily seen edema, minimally palpable, involving up to 1/3 of the treatment area Grade 3 = Moderate - easily seen edema and typically palpable, involving between 1/3 to 2/3 of the treatment area Grade 4 = Severe - easily seen edema, indurated in some areas, involving over 2/3 of the treatment area
Stinging/Burning | Baseline
  STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Stinging/Burning | Month 3
  STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Stinging/Burning | Month 6
  STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Stinging/Burning | Month 9
  STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Stinging/Burning | Month 12
  STINGING AND BURNING SCALE Grade 0 = None Grade 1 = Minimal, barely perceptible -tolerable and little discomfort Grade 2 = Moderate - tolerable, but causes some discomfort Grade 3 = Severe - very uncomfortable or intolerable
Scaling & Dryness | Baseline
  SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Scaling & Dryness | Month 3
  SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Scaling & Dryness | Month 6
  SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Scaling & Dryness | Month 9
  SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Scaling & Dryness | Month 12
  SCALING AND DRYNESS SCALE Grade 0 = None Grade 1 = Minimal - barely perceptible desquamation Grade 2 = Mild - limited areas of fine desquamation in up to 1/3 of the treatment area Grade 3 = Moderate - fine desquamation involving 1/3 to 2/3 of the treatment area or limited areas of coarser scaling Grade 4 = Severe - coarser scaling involving more than 2/3 of the treatment area or limited areas of very coarse scaling
Oozing/Vesiculation/Crusting | Baseline
  OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Oozing/Vesiculation/Crusting | Month 3
  OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Oozing/Vesiculation/Crusting | Month 6
  OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Oozing/Vesiculation/Crusting | Month 9
  OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above
Oozing/Vesiculation/Crusting | Month 12
  OOZING/VESICULATION/CRUSTING Grade 0 = None Grade 1 = Minimal - a single area of oozing, vesiculation or crusting 3 mm diameter or less in size Grade 2 = Mild - two to four areas of oozing, vesiculation or crusting 3 mm diameter or less in size OR a single area larger than 3 mm diameter in size Grade 3 = Moderate - more than a single area of oozing, vesiculation or crusting larger than 3 mm diameter in size or more than four areas of 3 mm diameter or less in size Grade 4 = Severe - any degree of oozing, vesiculation or crusting greater than (3) above

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Marcus, MD, PhD, Study Director — DUSA Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - UCSD Dermatology, San Diego, California
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - MOORE Clinical Research, Inc, Brandon, Florida
  - Spencer Clinical Services, St. Petersburg, Florida
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Shideler Clinical Research Center, Carmel, Indiana
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Oregon Dermatology and Research Center, Portland, Oregon
  - J&S Studies, Inc, College Station, Texas
  - Suzanne Bruce and Associates, P.A.,The Center for Skin Research, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia